CLINICAL TRIAL: NCT01603147
Title: A Phase Ia, Double-blind, Randomized, Placebo-controlled, Ascending IV Single-dose Study to Evaluate the Safety and Pharmacokinetics of ch mAb7F9 in Healthy Subjects
Brief Title: Safety Study of Ch-mAb7F9 for Methamphetamine Abuse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InterveXion Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXT TOA62936; R01DA031944 (NIH)
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Methamphetamine Abuse
Keywords: methamphetamine; monoclonal antibody
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): A total of 10 subjects will receive placebo
  Interventions: Biological: normal saline
- ch-mAb7F9 (Experimental): The single doses to be administered in each cohort are 0.2, 0.6, 2, 6, and 20 mg/kg, respectively.
  Interventions: Biological: ch-mAb7f9

INTERVENTIONS:
Biological: normal saline — saline 225 ml
  Arms: Saline
Biological: ch-mAb7f9 — The single doses to be administered in each cohort are 0.2, 0.6, 2, 6, and 20 mg/kg, respectively. Volume to be administered 225 ml
  Arms: ch-mAb7F9

SUMMARY:
The primary objective is to determine the safety and tolerability of single, ascending intravenous doses of ch-mAb7F9 in healthy subjects via physical examinations and adverse event, vital sign, electrocardiogram (ECG), and clinical laboratory testing.Phase 1a, randomized, placebo-controlled, first-in-human (FIH) study of intravenously administered ch-mAb7F9. The study will be a double-blind, dose-escalation study. Each subject will receive a single dose of ch-mAb7F9 or placebo (saline).

DETAILED DESCRIPTION:
There will be 5 dose groups. At the beginning of dosing in each group, 1 subject will receive the normal saline placebo and 1 will receive the active dose. The remainder of the dose group will receive their doses beginning 48 hr later, after safety evaluations. Dosing of the remaining subjects in each dose group will occur 1 at a time, with dosing in each subsequent subject separated by a minimum of 24 hr. Subsequent dose groups will receive their doses beginning approximately 2 weeks after dosing in the preceding group, pending safety analyses.

The single doses to be administered in each cohort are 0.2, 0.6, 2, 6, and 20 mg/kg, respectively. The starting dose will be 0.2 mg/kg, and the highest dose will be 20 mg/kg (up to a maximum of 1,500 mg), which is at least 20-fold lower than the no observable adverse effect level (NOAEL) in rats to ensure subject safety.

Ch-mAb7F9 will be administered intravenously (IV) with a saline flush to clear the administration tubing of residual ch-mAb7F9. Each dose of ch-mAb7F9 will be diluted in 225 ml of saline and given over two hours.

ELIGIBILITY:
Inclusion Criteria:

Subjects with the following criteria may be considered for inclusion in the study:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent form prior to performing any of the screening procedures.
2. Healthy, determined by the PI based on pre-study medical evaluation (medical history and physical examination, vital signs, ECG, and clinical laboratory evaluations).
3. Males or females between 18 to 50 years of age, inclusive.
4. The following applies to female subjects:

   - Nonchildbearing potential (surgically sterile [hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/occlusion] or post-menopausal 1 year with follicle stimulating hormone [FSH] > 40 U/L).

   OR

   - Nonpregnant, nonlactating females of childbearing age who agree to use medically acceptable forms of birth control (oral contraceptive pills; contraceptive patches; vaginal ring; diaphragm, sponge, or condom with spermicide; hormone injection; or intrauterine device) from screening to end of study follow-up, or whose partner has had a vasectomy.
5. The following applies to male subjects:

   * Need to have had a vasectomy or agree to use a condom and spermicide in addition to their female partners using a form of birth control.
   * Agree not to donate sperm for 90 days post dose.
6. Body mass index (BMI) between 18.5 and 30.5 kg/m2, inclusive, at screening. Body weight ≥ 50 kg and ≤ 100 kg at screening.
7. Nonsmokers or light smokers (< 10 cigarettes per day) able to refrain from smoking during the in-house period.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. A history of treatment with a monoclonal antibody in the past year,
2. likely allergy or sensitivity to ch-mAb7F9 based on known allergies to other mAbs, or which, in the opinion of the Principal Investigator (PI), suggests an increased potential for an adverse hypersensitivity to ch-mAb7F9,
3. a history of severe allergy (rash, hives, breathing difficulty, etc.) to any medications, either prescription or nonprescription, including dietary supplements or herbal medications,
4. a history of allergic or environmental bronchial asthma,
5. a clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, gastrointestinal, cardiovascular, pulmonary (including chronic asthma), endocrine (eg, diabetes), central nervous, or hematologic systems, or recent clinically significant surgery,
6. a history of seizure, epilepsy, severe head injury in the opinion of the PI, multiple sclerosis, or other known neurological conditions,
7. abnormal pre-admission vital signs, physical examination, clinical laboratory, or any safety variable which is considered clinically significant for this population by the PI or Sponsor (or designee), (volunteers who have or are suspected to have Gilbert's syndrome will be discussed on a case by case basis by the PI, Medical Monitor, and Sponsor),
8. a planned or scheduled surgical procedure during the study,
9. a clinically significant mental or physical illness within 1 year prior to the first dose, including a history of alcohol and/or drug abuse (DSM IV criteria) within 1 year prior to the first dose of study medication,
10. any history of stimulant use or abuse, including methamphetamine, amphetamine, or MDMA (ecstasy),
11. a recent (within 30 days of the first dose of study medication) donation of plasma or blood,
12. treatment with any medications, either prescription or nonprescription, including dietary supplements or herbal medications, within 14 days prior to the first dose of study medication (exceptions are nonprescription topical medications that are not systemically absorbed, acetaminophen, or vitamins at recommended daily doses),
13. ingestion of any known hepatic or renal clearance altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, St. John's Wort, etc.) within a period of 90 days prior to the first dose of study medication,
14. ingestion of any approved prescription anti-obesity drug or taken any over-the-counter medication for weight loss within a period of 90 days prior to the first dose of study medication,
15. ingestion or use of any investigational medication or device within 30 days prior to the first dose of study medication; ingestion or use of any investigational anti-obesity medication is prohibited within 3 months prior to the first dose of study medication,
16. acute illness within 5 days prior to the first dose of study medication, e.g., flu syndrome, gastrointestinal (GI) virus, or clinically significant indigestion (e.g., reflux) based on the discretion of the PI,
17. a positive test for HBsAG, Hepatitis C antibody, Hepatitis A IgM, or Human Immunodeficiency Virus (HIV) Viral Serology tests at the screening visit,
18. a positive urine alcohol test at screening or on Day -1; positive urine drug test for illicit substances (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, tetrahydrocannabinol [THC], phencyclidine, propoxyphene or MDMA) at screening or Day -1.
19. limited mental capacity to the extent that the subject cannot provide legal consent or understand information regarding the study,
20. a requirement for a special diet other than vegetarian or has a significant food allergy or intolerance,
21. any subject judged by the PI or Sponsor (or designee) to be inappropriate for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety | 21 weeks
  The primary outcome is to determine the safety and tolerability of single, ascending intravenous doses of ch-mAb7F9 in healthy subjects via physical examinations and adverse event, vital sign, electrocardiogram (ECG), and clinical laboratory testing.

SECONDARY OUTCOMES:
Pharmacokinetics | 21 weeks
  A secondary outcome is to characterize the pharmacokinetics of ch-mAb7F9 following single, ascending intravenous doses of ch-mAb7F9 in healthy subjects by measurement of mAb serum concentrations
Immunogenicity | 21 weeks
  A secondary outcome is to characterize the immune response following single, ascending intravenous doses of ch-mAb7F9 in healthy subjects by measurement of human anti-ch-mAb7F9 antibody (HACA) serum titers.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase 1 Services, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Harris AC, LeSage MG, Shelley D, Perry JL, Pentel PR, Owens SM. The anti-(+)-methamphetamine monoclonal antibody mAb7F9 attenuates acute (+)-methamphetamine effects on intracranial self-stimulation in rats. PLoS One. 2015 Mar 5;10(3):e0118787. doi: 10.1371/journal.pone.0118787. eCollection 2015. PMID 25742165